CLINICAL TRIAL: NCT01968135
Title: Does Concomitant Use of Combined Oral Hormonal Steroids Stop Bleeding in Women Using Etonogestrel Implants (Implanon/Nexplanon®)?: A Randomized Controlled Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-1702
Record Dates: First submitted 2013-10-18; First posted 2013-10-23 (Estimated); Results first posted 2016-05-05 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-04

CONDITIONS: Uterine Hemorrhage; Contraception
MeSH Terms: conditions — Uterine Hemorrhage | interventions — Contraceptives, Oral, Combined

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator): Placebo Sugar Pill
  Interventions: Drug: Placebo Sugar Pill
- Combined Oral Contraceptive Pill (Experimental): 150 mcg levonorgestrel and 30 mcg ethinyl estradiol combined oral contraceptive pill
  Interventions: Drug: Combined Oral Contraceptive Pill

INTERVENTIONS:
Drug: Combined Oral Contraceptive Pill — 150 mcg levonorgestrel and 30 mcg ethinyl estradiol combined oral contraceptive pill
  Arms: Combined Oral Contraceptive Pill
Drug: Placebo Sugar Pill — Placebo Sugar Pill
  Arms: Sugar Pill

SUMMARY:
The specific aims are to determine if more women using Etonogestrel (ENG) contraceptive implants who report a bleeding-spotting episode of at least seven days will stop bleeding within 3 days of beginning a 14-day course of combined oral hormonal steroids, as compared to women receiving 14 days of placebo.

DETAILED DESCRIPTION:
The ENG contraceptive implant (Implanon/Nexplanon®), is a silicone- free, single rod subdermal contraceptive implant that contains 68 mg of etonogestrel, is approved for use for three years, and is one of the most effective forms of contraception available (1). ENG contraceptive implants are easily inserted and removed (1,2), offer quick return to fertility (2), are cost-effective and cost-saving (3,4) and offer non-contraceptive benefits such as improvement in pain for patients with complaints of dysmenorrhea (5).

Hypothesis: Women using ENG contraceptive implants who report a bleeding-spotting episode of at least seven days will be more likely to stop bleeding within 3 days of beginning a 14-day course of combined oral hormonal steroids compared to women receiving 14 days of placebo.

ELIGIBILITY:
Inclusion Criteria:

* All female
* English or Spanish speaking women
* between the ages of 18-44
* using an ENG contraceptive implant who complain of bothersome bleeding and have a current bleeding episode of at least seven days will be invited to participate.

Exclusion Criteria:

* Category 3 or 4 contraindications to estrogen therapy according to the Centers for Disease Control 2010 Medical Eligibility Criteria.
* Category 3 contraindications: less than 1 month postpartum if breastfeeding, less than 21 days postpartum if not breastfeeding, history of Deep Vein Thrombosis (DVT) /Pulmonary Embolism (PE) not on anticoagulant therapy and no risk factors, Deep venous thrombosis/Pulmonary Embolus on established anticoagulant therapy and no risk factors, history of malabsorptive bariatric surgery, greater than or equal to months post peripartum cardiomyopathy with normal to mildly impaired cardiac function, greater than or equal to 35 years old with less than 15 cigarettes smoked per day, multiple risk factors for arterial cardiovascular disease, adequately controlled hypertension, blood pressure 140-159/90-99 mm Hg, migraines without aura less than 35 years old, past breast cancer and no evidence of recurrent disease for 5 years, diabetes with retinopathy, neuropathy, nephropathy (category 3 or 4 depending on severity), diabetes greater than 20 years duration or associated with other vascular disease, medically treated symptomatic gallbladder disease or current symptomatic gallbladder disease, past combined oral contraceptive pill related cholestasis, acute viral hepatitis, hepatocellular adenoma, hepatoma, use of ritonavir-boosted protease inhibitors, anticonvulsant therapy use including phenytoin, carbamazepine, barbiturates, primidone, topiramate, oxcarbazepine, and lamotrigine, use of Rifampicin,
* Category 4 contraindications: less than 6 months post peripartum cardiomyopathy with normal to mildly impaired cardiac function, any time following peripartum cardiomyopathy with moderately to severely impaired cardiac function, greater than or equal to 35 years old with greater than 15 cigarettes smoked per day, multiple risk factors for arterial cardiovascular disease, blood pressure greater than or equal to 160/100 mm Hg, high risk for recurrent DVT/PE, acute DVT/PE, DVT/PE and on established anticoagulant therapy with greater than or equal to 1 risk factor for recurrent DVT/PE, major surgery/prolonged immobilization, known thrombogenic mutations, current and history of ischemic heart disease, history of stroke, complicated valvular heart disease, systemic lupus erythematosus (SLE) with positive or unknown antiphospholipid antibodies, migraines without aura greater than or equal to 35 years old, migraines with aura at any age, current breast cancer, complicated solid organ transplantation
* Body mass index (BMI) greater than 35.
* A systolic blood pressure greater than 135 on more than 2 occasions. assuring the measurements are separated by an interval of at least 15 minutes.
* A diastolic blood pressure greater than 85 on more than 2 occasions. assuring the measurement are separated by an interval of at least 15 minutes.
* A positive pregnancy test.
* A positive chlamydia test.
* Unable or unwilling to swallow pills.
* A medical condition deemed severed by a physician investigator.
* A participant taking a liver enzyme inducing drug.
* A known allergy to levonorgestrel or ethinyl estradiol.
* An abnormal speculum exam (i.e. bleeding ectropion or cervical mass).
* Does not meet appropriate cervical cytology screening guidelines.
* Cervical procedure done in the past 3 months.
* On a concurrent hormonal contraceptive and unwilling to discontinue.
* Breast lesions

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Guiahi, MD, MSc, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Guiahi M, McBride M, Sheeder J, Teal S. Short-Term Treatment of Bothersome Bleeding for Etonogestrel Implant Users Using a 14-Day Oral Contraceptive Pill Regimen: A Randomized Controlled Trial. Obstet Gynecol. 2015 Sep;126(3):508-513. doi: 10.1097/AOG.0000000000000974. PMID 26181091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women were invited to participate after being seen at one of our institution's clinics with the complaint of bothersome bleeding during use of etonogestrel implant, or after responding to advertisements posted on the internet, in the local newspaper, or around public venues. Women were enrolled and followed from November 2013 - December 2014.
Pre-assignment Details: Interested women were screened by phone and subsequently invited for a screening visit. At this visit they were assessed for eligibility based on the specified inclusion/exclusion criteria.
Period: Overall Study
Arm/Group | Sugar Pill | Combined Oral Contraceptive Pill
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Combined Oral Contraceptive Pill | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (4.8) | 21.4 (3) | 21.9 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 12 | 10 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 13 | 12 | 25
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.2 (2.9) | 23.3 (3.5) | 23.2 (3.2)
Total days of current bleeding episode [Mean (Standard Deviation); unit: days] | 49.6 (44.6) | 30.3 (37.7) | 39.9 (41.8)

OUTCOME MEASURES:

1. Primary Outcome: Cessation of Vaginal Bleeding
Description: Proportion of women in each group who stopped bleeding during therapy and continued to report no bleeding at the end of the 14-day treatment period.
Time Frame: At day 3 of 14 day course of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Sugar Pill | Combined Oral Contraceptive Pill
Number analyzed (Participants) | 16 | 16
percentage of participants | 37.5 | 87.5

2. Secondary Outcome: Number of Days Until Temporary Interruption of Bleeding During Therapy Occurred
Time Frame: over the 14 day course of study drug
Measure: Median (Full Range); unit: days
Arm/Group | Sugar Pill | Combined Oral Contraceptive Pill
Number analyzed (Participants) | 16 | 16
days | 9 [5 to 14] | 5 [1 to 13]

3. Secondary Outcome: Number of Days Without Bleeding During Therapy
Time Frame: Over the 14 day course of study drug
Measure: Median (Full Range); unit: days
Arm/Group | Sugar Pill | Combined Oral Contraceptive Pill
Number analyzed (Participants) | 16 | 16
days | 3.5 [0 to 11] | 9 [1 to 13]

4. Secondary Outcome: Number of Days to Recurrence of Bleeding After Discontinuation of Therapy
Time Frame: Up to six months
Measure: Median (Full Range); unit: days
Arm/Group | Sugar Pill | Combined Oral Contraceptive Pill
Number analyzed (Participants) | 16 | 16
days | 10 [3 to 87] | 5.5 [1 to 131]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Sugar Pill | Combined Oral Contraceptive Pill
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No